CLINICAL TRIAL: NCT05097352
Title: Effects of a High-intensity Interval Training (HIIT) Exercise Intervention on Sleep in Women Exposed to Trauma: A Randomized Controlled Trial
Brief Title: Effects of a Short-term Exercise Intervention on Sleep in Women Exposed to Trauma: A Randomized Controlled Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Georgia (Other)
Responsible Party: Principal Investigator, Patrick O'Connor, Professor, University of Georgia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: PROJECT00004322
Record Dates: First submitted 2021-09-28; First posted 2021-10-28 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Traumatic Stress Disorder; Post Traumatic Stress Disorder; Trauma and Stressor Related Disorders; Mental Disorders; Exercise
MeSH Terms: conditions — Stress Disorders, Traumatic; Stress Disorders, Post-Traumatic; Trauma and Stressor Related Disorders; Mental Disorders; Motor Activity | interventions — High-Intensity Interval Training; Waiting Lists

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Interval Training (HIIT) (Experimental): High-intensity interval training will be performed three times a week for a total of six weeks.
  Interventions: Behavioral: High Intensity Interval Training (HIIT)
- Waitlist Control (Sham Comparator): Waitlist participants were tested on the outcomes at the same time points as the treatment group (i.e., HIIT). Following completion of the waitlist treatment, participants will be eligible to receive a supervised exercise program (no data will be collected). The waitlist participants formed a no-treatment control group.
  Interventions: Other: Waitlist

INTERVENTIONS:
Behavioral: High Intensity Interval Training (HIIT) — Twenty minutes of HIIT will be completed three days a week for six weeks.
  Arms: High Intensity Interval Training (HIIT)
Other: Waitlist — Waitlist participants will be tested on the outcomes at the same time points as the treatment group.
  Arms: Waitlist Control

SUMMARY:
This study aims to test whether sleep improvements, following 6 weeks of high-intensity interval training exercise among adult women exposed to a traumatic event, are mediated by improvements in heart rate variability or decreased anxiety and hyperarousal symptoms.

DETAILED DESCRIPTION:
A total of 60 women with below-average sleep quality and physical activity levels who also screen positive for PTSD on the Post-traumatic Diagnostic Scale (PDS-5) will be randomized to either six weeks of exercise training or a waitlist control. Twenty minutes of high intensity interval training will be performed three times per week for six-weeks. Heart rate variability will be measured at rest, during, and following a cognitive task. Psychometric measures supported by strong validity evidence will assess self-reported anxiety and PTSD symptoms, and sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* self-reported exposure to a traumatic event
* persistent (> 1 month) PTSD-related symptoms adequate to screen positive for PTSD or self-reported history of a prior PTSD diagnosed by a health care professional.
* poor sleep quality (Pittsburgh Sleep Quality Index >5)
* failure to meet recommended level of aerobic or resistance training during leisure time. Physical activity for U.S. adults (<150-mins of moderate or 75-mins of vigorous physical activity [or a combination] per week and/or < 2 days a week of resistance training targeting the major muscle groups).
* able to safely perform high-intensity exercise
* aged 18-39 years
* non-smoker
* willing to avoid alcohol and vigorous physical activity 24 hours before visiting the lab
* willing to avoid caffeine for 12 hours before visiting the lab

Exclusion Criteria:

* Pregnant, lactating, or plans to become pregnant over the next 2 months.
* Individuals who started taking medication for anxiety or depression-related symptoms within the last month.
* Individuals currently taking beta-blockers or other medications/substances (marijuana and other illegal drugs) that impact heart rate.
* History of reproductive disorders (e.g., premenstrual dysphoric disorder or polycystic ovary syndrome), cardiovascular (e.g., cardiac arrhythmia), or pulmonary disorders (e.g., asthma).
* Pain intensity of 8 or greater in the thigh or foot in the past month
* Probable alcohol use disorder

Ages: 18 Years to 39 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 41 (Actual)
Dates: Start 2022-01-24 (Actual); Primary Completion 2023-03-31 (Actual); Study Completion 2023-03-31 (Actual)

PRIMARY OUTCOMES:
Pittsburg Sleep Quality Index (PSQI) | Change from Baseline to week 7
  The PSQI consists of 19 items. Scores range from 0-21, higher scores indicate poorer sleep quality. A global score ≥5 indicates poor sleep quality.
Heart Rate Variability | Change from Baseline to Week 7
  High frequency (HF) and low frequency (LF) domains of heart rate variability will be assessed before, during, and following a cognitive task.
State Trait Anxiety Inventory (STAI-Y2) | Change from Baseline to Week 7
  The STAI-Y2 Trait subscale consists of 20-item and will assess anxiety. The total score ranges from 20-80; higher scores indicate greater trait anxiety.
The Posttraumatic Diagnostic Scale-5 (PDS-5) | Change from Baseline to Week 7
  The PDS-5 consists 24-item scale and will assess PTSD symptoms based on the diagnostic criteria for the DMS-5. The full PDS-5 assesses trauma history, symptom onset, and index of trauma. The total score ranges from 0-80.

CONTACTS AND LOCATIONS:
Overall Officials: Patrick J O'Connor, PhD, Principal Investigator — University of Georgia
Locations (1):
- University of Georgia, Athens, Georgia, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] McGranahan MJ, O'Connor PJ. Effect of high-intensity interval training exercise on sleep quality in women with probable post-traumatic stress disorder: A pilot randomized controlled trial. Sleep Med. 2025 May;129:245-256. doi: 10.1016/j.sleep.2025.02.029. Epub 2025 Feb 21. PMID 40056660

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT05097352/Prot_SAP_000.pdf
  • Informed Consent Form (2021-09-16): https://cdn.clinicaltrials.gov/large-docs/52/NCT05097352/ICF_001.pdf